CLINICAL TRIAL: NCT03773315
Title: Effect of Ulmus Macrocarpa Hance Extract on Lipid Profile in Adults With Dyslipidemia: a RCT
Brief Title: Ulmus Macrocarpa Hance Extract and Lipid Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sang Yeoup Lee (Other)
Responsible Party: Sponsor-Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Organization: Pusan National University Yangsan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2018-029
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UMH group (Experimental): This group takes UMH extract for 12 weeks
  Interventions: Dietary Supplement: UMH extract
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: UMH extract — Schisandra chinensis extract 500 mg/day for 12 weeks
  Arms: UMH group
Dietary Supplement: Placebo — Starch placebo 500 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the Ulmus Macrocarpa Hance extract on lipid profile in adults with dyslipidemia for 12 weeks.

DETAILED DESCRIPTION:
Previous another our study have indicated that Ulmus Macrocarpa Hance extract (UMH) may have the ability to decrease blood cholesterol. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the UMH on lipid profile in adults with dyslipidemia; the safety of the compound are also evaluate. The Investigators examine total cholesterol, HDL-cholesterol, triglyceridemia, LDL-cholesterol, and other biochemical parameters at baseline, as well as after 6 and 12 weeks of intervention. Eighty adults were administered either 500 mg of UMH or a placebo each day for 12 weeks;

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol ranging from 130 to 190 mg/dL

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 80 IU/L and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of ischemic heart disease or cerebrovascular disease
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 12 weeks
  LDL cholesterol

SECONDARY OUTCOMES:
Total cholesterol | 12 weeks
  Total cholesterol
Triglyceride | 12 weeks
  Triglyceride
HDL cholesterol | 12 weeks
  HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Integrated Research Institute for Natural Ingredients and Functional Foods, Yangsan, South Korea

REFERENCES:
- [Derived] Lee YL, Lee SY. Potential lipid-lowering effects of Ulmus macrocarpa Hance extract in adults with untreated high low-density lipoprotein cholesterol concentrations: A randomized double-blind placebo-controlled trial. Front Med (Lausanne). 2022 Nov 1;9:1000428. doi: 10.3389/fmed.2022.1000428. eCollection 2022. PMID 36388925